CLINICAL TRIAL: NCT01809990
Title: Internet-delivered Cognitive Behavior Therapy for Adolescents With Obsessive-Compulsive Disorder - a Pilot Study
Brief Title: Internet-delivered CBT for Adolescents With Obsessive-Compulsive Disorder - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eva Serlachius (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Sponsor-Investigator, Eva Serlachius, PhD, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIPOCD1
Record Dates: First submitted 2013-02-17; First posted 2013-03-13 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: cognitive behavior therapy; pediatric obsessive-compulsive disorder; internet-delivered cognitive behavior therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- internet-delivered cognitive behavior therapy (Experimental): Participants will be assigned to a 12 weeks internet-delivered cognitive behavior therapy program including therapist contact via an internet platform and telephone.
  Interventions: Behavioral: Internet-delivered Cognitive Behavior Therapy

INTERVENTIONS:
Behavioral: Internet-delivered Cognitive Behavior Therapy

SUMMARY:
The main goal of this trial is to study the feasibility and effectiveness of internet-delivered cognitive behavior therapy for adolescents with obsessive-compulsive disorder.

ELIGIBILITY:
Inclusion Criteria:

* a primary diagnosis of OCD as defined by DSM-IV TR
* a total score of above 15 on the CY-BOCS
* age between 12 and 17 years
* ability to read and write Swedish
* daily access to the internet
* a parent that is able to co-participate in the treatment
* Participants on psychotropic medication must have been on a stable dose for the last 6 weeks prior to baseline assessment
* signed informed consent

Exclusion Criteria:

* diagnosed autism spectrum disorder, psychosis or bipolar disorder
* suicidal ideation
* ongoing substance dependence
* subject not able to read or understand the basics of the ICBT self-help material
* completed CBT for OCD within last 12 months (defined as at least 5 sessions CBT including exposure and response prevention)
* ongoing psychological treatment for OCD or another anxiety disorder

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Children's Yale Brown Obsessive Compulsive Scale, CY-BOCS | Baseline, 12 weeks after treatment starts, 3 and 6 months after treatment has ended
  Change from Baseline of obsessions and compulsions after 12 weeks and at 3- and 6 months after treatment.

SECONDARY OUTCOMES:
Spence Child Anxiety Scale - Child and Parent version | Baseline, 12 weeks after treatment starts, 3 and 6 months after treatment has ended
  Spence Child Anxiety Scale - Child and Parent version (SCAS/P, Spence, 1998) will be used as a child and parent self-report measure of anxiety related psychopathology.
Child Depression Inventory | Baseline, 12 weeks after treatment starts, 3 and 6 months after treatment has ended
  Symptom severity of depression in the adolescent will be assessed with Child Depression Inventory (CDI, Kovacs, 1985).
Strengths Difficulties Questionnaire | Baseline, 12 weeks after treatment starts, 3 and 6 months after treatment has ended
  Strengths Difficulties Questionnaire (SDQ, Goodman, 1997) is a widely used self- and parent-report behavioral screening questionnaire with six subscales: emotional problems, conduct problems, hyperactivity-inattention, peer problems, prosocial behavior
Children's Obsessional Compulsive Inventory Revised | Baseline, 12 weeks after treatment starts, 3 and 6 months after treatment has ended
  The Children's Obsessional Compulsive Inventory Revised, (CHOCI-R, Shafran et al., 2003) is a self- and parent-report measure of pediatric OCD symptom severity.
Child Obsessive-Compulsive Impact Scale - Revised | Baseline, 12 weeks after treatment starts, 3 and 6 months after treatment has ended
  Child Obsessive-Compulsive Impact Scale - Revised (COIS-R, Piacentini, Peris, Bergman, Chang, & Jaffer, 2007) is a self- and parent-report scale of OCD symptom impact on everyday life.

OTHER OUTCOMES:
Patient Health Questionnaire PHQ-9 | Baseline, 12 weeks after treatment starts, 3 and 6 months after treatment has ended
  Patient Health Questionnaire PHQ-9 (Kroenke, Spitzer, & Williams, 2001) is a brief self-report measure of depressive symptoms in adults. PHQ-9 will be used to measure parental depressive symptoms.
GAD-7 | Baseline, 12 weeks after treatment starts, 3 and 6 months after treatment has ended
  GAD-7 (Spitzer, Kroenke, Williams, & Löwe, 2006) is a brief self-report measure of symptoms of general anxiety in adults. GAD-7 will be used to measure symptoms of anxiety in the parents.
Obsessive Compulsive Inventory - Revised | Baseline, 12 weeks after treatment starts, 3 and 6 months after treatment has ended
  Obsessive Compulsive Inventory - Revised (OCI-R, Foa et al., 2002) is a reliable and valid 18-item self-report scale for screening of OCD in adults and will be used to measure parental OC symptoms of both parents.
Family Accommodation Scale, Parent-Report | Baseline, 12 weeks after treatment starts, 3 and 6 months after treatment has ended
  Family Accommodation Scale, Parent-Report (FAS-PR, Flessner et al., 2009). The parent-report version of the FAS consists of 12 items focusing on accommodation behaviors of parents with a child with OCD.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Serlachius, PhD, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska insititute, Stockholm, Sweden

REFERENCES:
- [Background] Flessner CA, Sapyta J, Garcia A, Freeman JB, Franklin ME, Foa E, March J. Examining the Psychometric Properties of the Family Accommodation Scale-Parent-Report (FAS-PR). J Psychopathol Behav Assess. 2009 Mar;31(1):38-46. doi: 10.1007/s10862-010-9196-3. PMID 21743772
- [Background] Foa EB, Huppert JD, Leiberg S, Langner R, Kichic R, Hajcak G, Salkovskis PM. The Obsessive-Compulsive Inventory: development and validation of a short version. Psychol Assess. 2002 Dec;14(4):485-96. PMID 12501574
- [Background] Goodman R. The Strengths and Difficulties Questionnaire: a research note. J Child Psychol Psychiatry. 1997 Jul;38(5):581-6. doi: 10.1111/j.1469-7610.1997.tb01545.x. PMID 9255702
- [Background] Kovacs M. The Children's Depression, Inventory (CDI). Psychopharmacol Bull. 1985;21(4):995-8. No abstract available. PMID 4089116
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Piacentini J, Peris TS, Bergman RL, Chang S, Jaffer M. Functional impairment in childhood OCD: development and psychometrics properties of the Child Obsessive-Compulsive Impact Scale-Revised (COIS-R). J Clin Child Adolesc Psychol. 2007 Oct-Dec;36(4):645-53. doi: 10.1080/15374410701662790. PMID 18088221
- [Background] Scahill L, Riddle MA, McSwiggin-Hardin M, Ort SI, King RA, Goodman WK, Cicchetti D, Leckman JF. Children's Yale-Brown Obsessive Compulsive Scale: reliability and validity. J Am Acad Child Adolesc Psychiatry. 1997 Jun;36(6):844-52. doi: 10.1097/00004583-199706000-00023. PMID 9183141
- [Background] Shafran R, Frampton I, Heyman I, Reynolds M, Teachman B, Rachman S. The preliminary development of a new self-report measure for OCD in young people. J Adolesc. 2003 Feb;26(1):137-42. doi: 10.1016/s0140-1971(02)00083-0. PMID 12550826
- [Background] Spence SH. A measure of anxiety symptoms among children. Behav Res Ther. 1998 May;36(5):545-66. doi: 10.1016/s0005-7967(98)00034-5. PMID 9648330
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Derived] Lenhard F, Vigerland S, Andersson E, Ruck C, Mataix-Cols D, Thulin U, Ljotsson B, Serlachius E. Internet-delivered cognitive behavior therapy for adolescents with obsessive-compulsive disorder: an open trial. PLoS One. 2014 Jun 20;9(6):e100773. doi: 10.1371/journal.pone.0100773. eCollection 2014. PMID 24949622